CLINICAL TRIAL: NCT00929565
Title: Utility of Serum and Bronchoalveolar Fluid Urokinase Like Plasminogen Activator Levels in Defining Patients at Higher Risk of Hemoptysis.
Brief Title: Urokinase Like Plasminogen Activator Levels in Patients Undergoing Bronchoscopy
Status: Completed | Type: Observational
Sponsor: University of Oklahoma (Other)
Responsible Party: Principal Investigator, Gary Kinasewitz, Principal Investigator, University of Oklahoma
Other Study IDs: 14455
Record Dates: First submitted 2009-06-24; First posted 2009-06-29 (Estimated); Last update posted 2012-04-09 (Estimated); Status verified 2012-04

CONDITIONS: Hemoptysis
Keywords: hemoptysis
MeSH Terms: conditions — Hemoptysis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Lung cancer: Comparison between individuals with and without pulmonary malignancy

SUMMARY:
Some of the risk factors for bleeding following bronchoscopy is having a malignancy or an immunocompromised state. The etiology of this remains uncertain. The investigators suspect that individuals with malignancy have abnormalities involving certain factors that influence the coagulation pathway.

The investigators plan to measure these factors prior to and after bronchoscopy.

DETAILED DESCRIPTION:
This is a prospective observational study looking at some coagulation factors in individuals with lung cancer. We are looking at BAL and plasma. We would like to see if there is a difference in the levels and if this is the reason behind the higher incidence of hemoptysis in patients with lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* Any patient scheduled to undergo bronchoscopy

Exclusion Criteria:

* Patients with evidence of coagulopathy either iatrogenic or the result of disease process - coagulopathy defined as elevated prothrombin time, activated partial thromboplastin time or platelet count less than 100,000
* Patients not scheduled to undergo bronchoalveolar lavage (BAL)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients from the VAMC in Oklahoma city
Sampling Method: Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2009-06; Primary Completion 2010-06 (Actual); Study Completion 2011-10 (Actual)

SECONDARY OUTCOMES:
Volume of blood loss during the procedure | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Jijo John, MD, Principal Investigator — University of Oklahoma
Locations (1):
- VA Medical Center, Oklahoma City, Oklahoma, United States